CLINICAL TRIAL: NCT05272371
Title: Immunotherapy With Dinutuximab Beta in Combination With Chemotherapy for the Treatment of Patients With Primary Neuroblastoma Refractory to Standard Therapy and With Relapsed or Progressive Disease
Acronym: ChIm-NB-PL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Walentyna Balwierz, Prof., Jagiellonian University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChIm-NB-PL
Record Dates: First submitted 2022-03-01; First posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: High-Risk Neuroblastoma
Keywords: neuroblastoma dinutuksymab beta chemoimmunotherapy
MeSH Terms: interventions — dinutuximab; Drug Therapy

STUDY DESIGN:
Intervention Model Description: Treatment group compared to historical group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Chemoimmunotherapy arm.
  Interventions: Combination Product: Chemoimmunotherapy (Dinutuximab beta in combination with chemotherapy)

INTERVENTIONS:
Combination Product: Chemoimmunotherapy (Dinutuximab beta in combination with chemotherapy) — Dinutuximab beta in combination with chemotherapy.

SUMMARY:
Safety evaluation and initial efficacy evaluation will be conducted in a group of patients as a non-commercial, open-label clinical trial of dinutuximab beta (Qarziba) phase IIa.

The investigational medicinal product will be dinutuximab beta (anti-GD2 antibodies against GD2 disialoganglioside on NBL cells) at a dose of 10 mg / m2 / day by continuous infusion for 5 days in combination with irinotecan / temozolomide, topotecan / temozolomide or N5 / N6 chemotherapy GPOH protocol.

The study group will be patients with recurrent / progression of NBL or disease resistant to first-line treatment, for whom there are currently no standards of management, and the treatment methods used so far do not give a chance to achieve a permanent remission of the disease. After diagnosis of relapse / progression or resistance to treatment, it is permissible to administer 2 cycles of standard chemotherapy prior to enrollment in the study.

The study plans to recruit 20 patients who will receive 5-7 cycles of DB with chemotherapy. The choice of an appropriate chemotherapy regimen will depend on the patient's prior treatment and tolerance.

The safety assessment will be conducted based on the registration of the types and frequency of adverse reactions identified on the basis of the registration of clinical parameters, symptoms and / or diseases reported by the patient or identified during the intervention and / or follow-up visits, abnormal laboratory and / or imaging test results.

The initial assessment of the effectiveness will consist in comparing the percentage of objective responses obtained and the annual EFS and PFS (imaging tests, including scintigraphy, bone marrow examination and tumor markers). The study also included an exploratory evaluation of the usefulness of immunological, genetic and other studies.

DETAILED DESCRIPTION:
Neuroblastoma (NBL) accounts for 8-10% of all childhood malignancies. It is the most common solid tumor outside the central nervous system in people <18 years of age. It occurs in 6-11 / 1 million children annually. In Poland, NBL is diagnosed annually in 60-70 patients, in 1/3 high-risk disease (HR). In 90% of children, NBL is diagnosed before the age of 5. The diagnosis is made on the basis of the histopathological assessment of the tumor tissue or the presence of NBL cells in the bone marrow together with elevated levels of catecholamines or their metabolites in the urine. The prognostic factors include the patient's age at diagnosis, stage of disease, tumor histopathology, DNA ploidy, MYCN gene status, chromosomal changes, and initial response to therapy. Due to the different course of the disease, the therapeutic decision is made after determining the risk group based on international criteria (International Neuroblastoma Risk Group Stage System, INRGSS and International Neuroblastoma Staging System, INSS). In the lowest-risk group, management is limited to observation or surgery, and in the intermediate-risk group, only standard low- and intermediate-intensity chemotherapy or combined with radiation therapy and surgery is performed. In contrast, HR-NBL uses intensive combination therapy, including standard induction chemotherapy, surgery, high-dose chemotherapy (HD-CHT) and autologous hematopoietic stem cell transplantation (auto-HSCT), radiotherapy and maintenance therapy with 13-cis retinoic acid and targeted immunotherapy with anti-GD2 antibodies. Treatment outcomes in NBL vary from spontaneous tumor regression in some infants to an OS rate of <50% despite intensive combination therapy in the HR-NBL group.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of NBL according to international criteria (International Neuroblastoma Risk Group, INRG).
2. Patients 1-18 years of age with HR-NBL with primary refractory disease, disease progression or recurrence.
3. Adequate function of vital organs (if abnormal, dysfunction below grade 4 according to the CTC AE WHO classification, except for disorders defined in the exclusion criteria).
4. Life expectancy ≥6 months.
5. Obtaining the informed written consent of the patient and/or statutory representative for the treatment.
6. Female patients of childbearing potential must consent to the use of effective contraception; Breastfeeding patients must consent to the termination of breastfeeding.
7. Patients who have previously received immunotherapy with DB or other anti-GD2 specific antibodies may be eligible for this study.

Exclusion Criteria:

1. Patients with toxicities of ≥3 CTCAE WHO grade, except hearing impairment, hematological disorders, liver and kidney disorders.
2. Patients with neurological toxicities of ≥2 CTCAE WHO grade.
3. Active life-threatening infection until stabilization of the patient's condition.
4. Pregnancy and / or lactation.
5. Sexually active patients who refuse to use an effective method of contraception.
6. Current treatment with experimental drugs or use of such treatment within 2 weeks before signing the informed consent to participate in the study.
7. Radiotherapy within 3 weeks prior to the start of the study.
8. Participation in another clinical trial within 6 months before signing the informed consent to participate in the trial (not applicable to clinical trials in 1st line of treatment in HR-NBL).
9. Lack of informed written consent to treatment.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of cycles aborted due to toxicity. | 12 months after end of treatment.
Number of cycles in which treatment interruptions due to the occurrence of side effects will be longer than provided for in the treatment protocol. | 12 months after end of treatment.
Number of episodes of Capillary Leak Syndrome, regardless of severity. | 12 months after end of treatment.
Number of episodes of cytokine release syndrome, regardless of severity. | 12 months after end of treatment.
Number of episodes of allergic reactions in CTCAE grade 3 and 4 (version in force at that time). | 12 months after end of treatment.
Number of hematological toxicities in grade 3 and 4 CTCAE (version in force at that time). | 12 months after end of treatment.
Number of neurological toxicity episodes, regardless of severity. | 12 months after end of treatment.
The percentage of patients with pupil disorders and / or visual disturbances. | 12 months after end of treatment.
Proportion of patients with renal or hepatic impairment in CTCAE grade 3 and 4 (version in force at that time). | 12 months after end of treatment.
Other side effects in grade 3 and 4 CTCAE (version in force at the time)3 and 4 (version in force at that time). | 12 months after end of treatment.

SECONDARY OUTCOMES:
Percentage of patients with complete remission assessed during the study and at the last visit. | 12 months after end of treatment.
Percentage of patients with partial remission assessed during the study and at the last visit. | 12 months after end of treatment.
Percentage of patients with disease stabilization assessed during the examination and at the last visit. | 12 months after end of treatment.
Percentage of patients PFS assessed during the study. | 12 months after end of treatment.
Percentage of patients ESF assessed during the study. | 12 months after end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Walentyna Balwierz, Prof., Principal Investigator — Jagiellonian University
Locations (1):
- University Children Hospital, Krakow, Malopolska, Poland

IPD SHARING:
Plan to Share IPD: Undecided